CLINICAL TRIAL: NCT06414863
Title: Treatment Effects of Invisalign Palatal Expander System and Hyrax Palatal Expander - A Randomized Controlled Trial
Brief Title: Effects of Invisalign Palatal Expander System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Principal Investigator, Heeyeon Suh, Assistant professor, University of the Pacific
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-43
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Palatal Expansion Technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Invisalign® Palatal Expander System (Experimental): Invisalign® Palatal Expander System will be delivered.
  Interventions: Device: IPE
- Hyrax-type maxillary expander (Active Comparator): Hyrax-type maxillary expander will be delivered. The Hyrax-type maxillary expander will include a midline self-locking screw, which is connected to the conventional molar bands or printed clasps, which are cemented on the maxillary first molars (or on the maxillary primary second molars), via 0.9 mm stainless-steel wire. The framework is soldered to the bands and extends on the palatal side to the primary canines or canines. The expander will be fabricated by a qualified laboratory technician
  Interventions: Device: HE

INTERVENTIONS:
Device: IPE — Invisalign palatal expander system:
  The Invisalign® Palatal Expander System (AlignTechnology, inc.) is 3D-printed orthodontic device for maxillary expansion.
  Arms: Invisalign® Palatal Expander System
Device: HE — Hyrax expander:
  The Hyrax-type maxillary expander will include a midline self-locking screw. The expansion screw is connected to the conventional molar bands or printed clasps, which are cemented on the maxillary first molars (or on the maxillary primary second molars), via 0.9 mm stainless-steel wire. The framework is soldered to the bands and extends on the palatal side to the primary canines or canines. The expander will be fabricated by a qualified laboratory technician
  Arms: Hyrax-type maxillary expander

SUMMARY:
The aim of this study is to evaluate the effectiveness of Invisalign Palatal Expander system ingrowing patients. This study compares the treatment outcomes of Invisalign Palatal Expander system to conventional treatments through randomized controlled trial.

ELIGIBILITY:
Inclusion criteria:

1. Mixed dentition phase with at least three nonmobile (stable) teeth which have more than 1/4 of primary molar root length left16 in either side
2. Early permanent dentition stage and early permanent dentition but second permanent molars not yet fully erupted in the arch
3. Unilateral or bilateral posterior cross bite patients; or Patients who have been diagnosed with transverse maxillary deficiency (Skeletal transverse discrepancy measured from the estimated center of resistances of the first molars17 ≤ - 3 mm);
4. Patients with Class I or Class II skeletal relationship
5. Subjects willing to consent to the trial

Exclusion Criteria:

1. Any general medical health problems which may influence treatment
2. Any craniofacial anomalies
3. Skeletal Class III patients
4. Mixed dentition patients with more than 2 heavily restored primary second or permanent first molars.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2028-05-10 (Estimated); Study Completion 2034-05-10 (Estimated)

PRIMARY OUTCOMES:
Width change | 12-18 months
  Transverse changes on CBCTs
Arch width change | 12-18 months
  Arch width change measured on digital study casts

SECONDARY OUTCOMES:
Cephalometric changes | 12-18 months
  Common Cephalometric measurements changes on CBCT analysis

CONTACTS AND LOCATIONS:
Overall Officials: Heeyeon Suh, Principal Investigator — University of the Pacific
Locations (1):
- University of the Pacific, San Francisco, California, United States